CLINICAL TRIAL: NCT01474161
Title: Comparative Bioavailability Study of a New GFT505 Formulation With the Existing One After 120 mg Single Oral GFT505 Administration and Assessment of the Gender Effect in Young Healthy Male and Female Volunteers Followed by a Single and Multiple Ascending Dose Safety, Tolerability and Pharmacokinetic Study of GFT505 in Overweight or Obese Subjects and in Diabetic Patients
Brief Title: Comparative Bioavailability - Gender Effect - Single and Multiple Ascending Dose Safety and Pharmacokinetic Study of GFT505
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genfit (Industry)
Collaborators: SGS Aster S.A.S. (Unknown); Naturalpha (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GFT505-111-7; 2011-004723-13 (EudraCT Number)
Record Dates: First submitted 2011-11-15; First posted 2011-11-18 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Type 2 Diabetes; Diabetes Mellitus, Type 2; Metabolic Diseases; Cardiovascular Diseases; Obese; Dyslipidemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Diseases; Cardiovascular Diseases; Obesity; Dyslipidemias | interventions — 2-(2,6-dimethyl-4-(3-(4-(methylthio)phenyl)-3-oxo-1-propenyl)phenoxyl)-2-methylpropanoic acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Matching placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- GFT505 20mg - old formulation (Active Comparator): Study Part I : dose level = 120mg
  Interventions: Drug: GFT505 120mg - old formulation
- GFT505 60mg - new formulation (Experimental): Study Part I : dose level = 120mg ; Study Part II : dose level = 180mg, 240mg and 300mg ; Study Part III : dose level = 120mg, 180mg and 240mg ; Study Part IV : dose level = 120mg or 180mg.
  Interventions: Drug: GFT505 120mg - new formulation; Drug: GFT505 180mg - new formulation; Drug: GFT505 240mg - new formulation; Drug: GFT505 300mg - new formulation

INTERVENTIONS:
Drug: GFT505 120mg - old formulation — hard gelatin capsules dosed at 60mg, one single oral administration (Study part I), 6 capsules with 250mL of water.
  Arms: GFT505 20mg - old formulation
Drug: GFT505 120mg - new formulation — hard gelatin capsules dosed at 60mg, one single oral administration (Study Part I) or multiple dose administration from Day 1 to Day 14 (Study Part III and IV), 2 capsules with 250mL of water.
  Arms: GFT505 60mg - new formulation
Drug: GFT505 180mg - new formulation — hard gelatin capsules dosed at 60mg, one single oral administration (Study Part II) or multiple dose administration from Day 1 to Day 14 (Study Part III and IV), 3 capsules with 250mL of water.
  Arms: GFT505 60mg - new formulation
Drug: GFT505 240mg - new formulation — hard gelatin capsules dosed at 60mg, one single oral administration (Study Part II) or multiple dose administration from Day 1 to Day 14 (Study Part III), 4 capsules with 250mL of water.
  Arms: GFT505 60mg - new formulation
Drug: GFT505 300mg - new formulation — hard gelatin capsules dosed at 60mg, one single oral administration (Study Part II), 5 capsules with 250mL of water.
  Arms: GFT505 60mg - new formulation
Drug: Placebo — hard gelatin capsules, one single oral administration (3 to 5 capsules with 250mL of water for Study Part II) or multiple dose administration from Day 1 to Day 14 (2 to 4 capsules with 250mL of water for Study Part III).
  Arms: Matching placebo

SUMMARY:
The Sponsor, Genfit, has developed a new formulation of GFT505 (60 mg). The objective is to compare the relative bioavailability between the new GFT505 formulation (capsule dosed at 60 mg GFT505) and the old GFT505 formulation (capsule dosed at 20 mg GFT505) in healthy male subjects and to assess the impact of gender on this relative bioavailability after administration in male and female subjects.

Using the new formulation, a single and a multiple ascending dose study will be performed in overweight or obese male subjects otherwise healthy whose demographic and physiological characteristics are thought to be closer to those of the target population (Type 2 diabetes). Thereafter, a group of male and female patients with Type 2 diabetes will receive multiple dose administration of GFT505.

DETAILED DESCRIPTION:
The study will be divided in 4 successive parts :

* Study Part I will be a comparative bioavailability between a new GFT505 formulation (capsule dosed at 60 mg GFT505 by capsule) and the old GFT505 formulation (capsule dosed at 20 mg GFT505 by capsule) coupled with an evaluation of the gender effect assessed with the new formulation. In this purpose a group of 12 male subjects will receive successively both formulations on a unique occasion in a randomized manner while a group of 12 female subjects will receive the new formulation on one occasion only. This part of the study will be done in healthy volunteers.
* Study Part II will be a single ascending dose to be run at a maximum of 3 dose levels. Subjects included in this part of the study will receive only one dose level to limit the exposure to GFT505. Three cohorts of 8 subjects are planned to be included. This part will be run in overweight or obese subjects.
* Study Part III will start after completion of the first Cohort of Study Part II. Study Part III will be a multiple ascending dose to be run at a maximum of 3 dose levels. Subjects included in this part of the study will receive only one dose level to limit the exposure to GFT505. Three cohorts of 12 subjects are planned to be included. This part will be run in overweight or obese subjects.
* Study Part IV will follow the same design and same treatment schedule than Study Part III but will be performed in the target population, patients with Type 2 diabetes and only one dose will be tested in study part IV.

ELIGIBILITY:
Inclusion Criteria:

Part I :

* Male or female healthy volunteers 18 to 45 years of age (inclusive).
* Subjects with a body mass index (BMI) ≥ 18 and ≤ 28 kg/m2 at screening.
* For female subjects of childbearing potential, use of double contraception method.
* Normal arterial blood pressure (BP) and pulse rate or, if abnormal, considered not clinically significant by the principal Investigator.

Part II and III :

* Male healthy volunteers 18 to 55 years of age (inclusive).
* Subjects with a BMI >28 and <35 kg/m2 at screening.
* Normal arterial BP and pulse rate or, if abnormal, considered not clinically significant by the principal Investigator.

Part IV :

* Male or female Type 2 diabetic patients 18 to 60 years of age.
* Females participating in the study must be either of non-child bearing potential or using an efficient double contraception.
* Currently treated with any antidiabetic treatment (a maximum of two anti-diabetic drugs including metformin in all cases) with the exception of insulin or GLP analogs and agonists therapy.
* Stable diabetes with glycosylated hemoglobin (HbA1c) < or =10% or less.
* Normal renal function as defined by a creatine clearance >90 mL/min calculated with the Cockcroft-Gault formula.
* Subjects with a BMI from 18 to 32 kg/m2 at screening.

Exclusion Criteria:

Part I :

* Who previously received GFT505.
* With any clinically significant abnormality following review of prestudy laboratory tests (Aspartate and Alanine aminotransferase must be within normal ranges), vital signs, full physical examination and Electrocardiogram.
* Who have a positive laboratory test for Hepatitis B surface antigen (HbsAg), or anti-HIV 1/2 (Human immunodeficiency virus) or anti-HCV (Hepatitis C virus) antibodies.
* Who are known or suspected alcohol or drug abusers (more than 14 units of alcohol per week, one unit = 8 g or about 10 mL of pure alcohol).
* Who drink more than 8 cups daily of beverage containing caffeine.
* Who have a positive laboratory test for urine drug screening (opiates, cocaine, amphetamine, cannabis, benzodiazepines).
* Who have undergone surgery or have donated blood within 12 weeks prior to the start of the study.
* Who have taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 2 weeks prior to the first dose administration.

Part II and III : specific additional exclusion criteria

- Who have taken fibrates within 6 weeks prior to the first dose administration.

Part IV : specific additional exclusion criteria

* With unstable proliferative retinopathy, macular oedema (fundus examination performed in the previous year will be considered relevant on Investigator's judgement).
* Who have taken fibrates within 6 weeks prior to the first dose administration.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters (Study Part I) | 24h post-dose
  For each subject at each Treatment Period, blood will be collected at the following time points: pre-dose, and 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 h post-dose.
Safety parameters (Study Parts II, III and IV) | Part II : 5 days ; Part III : 20 days ; Part IV : 20 days
  Monitoring for the occurrence of AEs. Changes in physical examination, vital signs (blood pressure and pulse rate), ECG, and clinical laboratory tests (biochemistry, hematology, and urinalysis).

SECONDARY OUTCOMES:
Safety parameters (Study Part I) | 12 days for male and 5 days for female
  Monitoring for the occurrence of AEs. Changes in physical examination, vital signs (blood pressure and pulse rate), ECG, and clinical laboratory tests (biochemistry, hematology, and urinalysis).
Pharmacokinetics parameters (Study Parts II, III and IV) | Part II : 24h post-dose ; Part III : 15 days ; Part IV : 15 days
  Study Part II : For each subject of each dose level, blood will be collected at the following time points: pre-dose, and 0.5, 1, 1.5, 2, 4, 6, 8, 12 and 24 h post-dose.
  Study Part III and Study Part IV : Assuming a once daily administration, blood will be collected at the following time points:
  * Day 1 pre-dose and 0.5, 1, 1.5, 2, 4, 6, 8, 12, and 24 h post-dose.
  * Days 3, 7, 10, 11, 12 and 13 pre-dose.
  * Day 14 pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, and 24 h post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Rémy Hanf, Development Director, Study Director — GENFIT, France; Philippe Betting, MD, Principal Investigator — SGS Aster S.A.S., Phase I Clinical Unit, France
Locations (1):
- SGS Aster S.A.S. - Phase I Clinical Unit, Paris, France